CLINICAL TRIAL: NCT07082712
Title: Study Of Thyroid Disorders In Patients With Acute Coronary Syndrome At Sohag University Hospitals .
Brief Title: Investigate Relationship Between Thyroid Disorders and Acute Coronary Syndrome.
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Abobakr, Resident doctor, Sohag University
Other Study IDs: Soh-Med--25-6-4MS
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Disorders With Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thyroid profile — Thyroid profile in patients with acute coronary syndrome within 24 hour from admission

SUMMARY:
Study Of Thyroid Disorders In Patients With Acute Coronary Syndrome At Sohag University Hospitals.

DETAILED DESCRIPTION:
Our aim of the study to investigate relationship between thyroid disorders and acute coronary syndrome .We will study 300 hospitalized patients with a diagnosis of ACS to determine the prevalence of thyroid disorders, and their relationship with other known coronary risk factors. All patients included in the study will be subjected to:

Detailed medical history Detailed clinical examination

Laboratory investigation:

Thyroid function Tests (TSH, FT3, FT4) will collect from all the patients within 24 h of their admission to the coronary care unit (CCU).

Serum lipogram. cardiac enzymes.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 20 years old who were diagnosed with ACS.

Exclusion Criteria: - Patients known hypothyroidism or hyperthyroidism on treatment. Patients presented by acute decompensated heart failure. Patients with advanced malignancies. Patients with acute pulmonary thromboembolism.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients With Acute Coronary Syndrome
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Thyroid disorders in patient with acute coronary syndrome | Baseline(6 months of start of research)
  Detection of Thyroid profile Tsh(µIU/mL))normal rang(.4-5.5). FreeT4(ng/dL) FreeT3(pmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa AbuBakr "MohamedAl-Mobdy", Study Chair — Shoag University Hospitals; Asmaa AbuBakr "MohamedAl-Mobdy ", Principal Investigator — Tertiary hospital
Locations (1):
- Faculty of medicine sohag University, Sohag, Egypt